CLINICAL TRIAL: NCT05869253
Title: The Efficacy of Attention Skill Therapy (ASTride), an Equine Assisted Occupational Therapy Intervention, for Children With Attention Deficit Hyperactivity Disorder (ADHD) on Cognitive-emotional Aspects, Daily Function and Participation
Brief Title: The Efficacy of Equine Assisted Occupational Therapy for Children With Attention Deficit Hyperactivity Disorder (ADHD) on Cognitive-emotional Aspects, Daily Function and Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Orit Bart PhD, Lead investigator, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003949-2
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Attention-deficit Hyperactivity Disorder
Keywords: Equine Assisted Occupational Therapy; ADHD; strategy based; Equine Assisted Services; horse therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: A prospective cohort study with Interrupted Time-Series design will be conducted.
Masking Description: The intervention will be administered by a licensed EAOT, and assessments will be done by a blinded licensed occupational therapist (OT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- children diagnosed with ADHD (Experimental): After completing an eligibility assessment, adequate participants will go through baseline assessment and 12 weeks of waiting without receiving intervention; b) pre-test, before first treatment session, end of 12 week waiting period; c) post-test after 12 weeks of intervention; d) post intervention assessment, three months follow up
  Interventions: Behavioral: The efficacy of Equine Assisted Occupational Therapy, for children with Attention Deficit Hyperactivity Disorder (ADHD) on cognitive-emotional aspects, daily function and participation

INTERVENTIONS:
Behavioral: The efficacy of Equine Assisted Occupational Therapy, for children with Attention Deficit Hyperactivity Disorder (ADHD) on cognitive-emotional aspects, daily function and participation — : A prospective cohort study with Interrupted Time-Series design will be conducted. Forty participants and their parents who were referred to EAOT will be recruited from the waiting list of Harey Yehuda stables. Assessments will take place at four time points. Time 1: baseline-when referred for EAOT. Time 2: pre-test, before first treatment session, end of 12 week waiting period. Time 3: post-test after 12 weeks of intervention and time 4: post intervention assessment, three months follow up. The intervention will be administered by a licensed EAOT, and assessments will be done by a blinded licensed occupational therapist (OT). Standardized assessment measures will be used to measure EFs, cognitive-emotional and sensory-motor aspects as well as participation at each time point.
  Other Names: Taking the Reins

SUMMARY:
The goal of this clinical trial is to develop and validate an Equine Assisted Occupational Therapy Intervention for children aged 6-12 with Attention Deficit Hyperactivity Disorder.

The research aims to study the effect of an EAOT intervention on cognitive-emotional aspects, daily function and participation among these children using various measurements including physiological measures (EEG, heart rate for rider and horse), questionnaires and different tasks. It aims to enable the creation of an evidence based protocol for professionals in order to provide a better suited therapy for children with ADHD and enable them to live a full life. Participants will enroll in a 12 week EAOT intervention including one session per week of 45 minutes with a waiting period prior the intervention. Participants will go through assessments prior waiting time, prior the intervention and post intervention.

DETAILED DESCRIPTION:
Introduction: Attention deficit/hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is currently one of the most common diagnoses given to children. ADHD is characterized by a developmental and chronic impairment, Executive Functions (EFs), cognitive-emotional and sensory-motor functions, as well as a wide variety of difficulties in daily tasks beyond the core symptoms. Literature review indicated that current intervention protocols include pharmacological treatment and address specific aspects such as behavioral or psychological, though scarce interventions address both.

Objectives: The purpose of this study is to examine the feasibility of conducting an Equine Assisted Occupational Therapy (EAOT) intervention for children with ADHD aiming to improve EFs, cognitive-emotional functions and participation.

Method: A prospective cohort study with Interrupted Time-Series design will be conducted. Forty participants and their parents who were referred to EAOT will be recruited from the waiting list of Harey Yehuda stables. Assessments will take place at four time points. Time 1: baseline-when referred for EAOT. Time 2: pre-test, before first treatment session, end of 12 week waiting period. Time 3: post-test after 12 weeks of intervention and time 4: post intervention assessment, three months follow up. The intervention will be administered by a licensed EAOT, and assessments will be done by a blinded licensed occupational therapist (OT). Standardized assessment measures will be used to measure EFs, cognitive-emotional and sensory-motor aspects as well as participation at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 12 years of age
* Diagnosis of ADHD from a medical professional based on DSM-5 criteria with or without medication (e.g., psychostimulant medication)
* General doctors' approval and referral for participating in EAS

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Neurological disorders (e.g., epilepsy)
* Children with additional developmental disorders (e.g., Autism, Cerebral Palsy)
* Children who will begin new medicine treatment or change existing treatment during intervention
* Children with severe sensory loss (e.g., blindness).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The Behavior Rating Inventory of Executive Function (BRIEF) (Gioia, Isquith, Guy, & Kenworthy, 2000) | 3 months
  standardized ecological rating scale filled by a parent, designed to reflect the neuropsychological constructs of EF in everyday situations for children aged 5-18

SECONDARY OUTCOMES:
the Tower of Hanoi test (Lezak et al., 2004). | 3 months
  The TOH test measures EF with non-verbal content and requires spatial perception of position. It requires a generation of a multistep sequence of move and strategy selection. It requires executing the sequence of moves while inhibiting the incorrect moves
The Brain Engagement Index; BEI (Shahaf et al., 2018) | 3 months
  a real-time electrophysiological marker for sustained attention extracted from a simple and easy-to-use one-channel NeuroSky EEG MindWave system
The new General Self-efficacy Scale (NGSE) | 3 months
  a 11-item questionnaire designed to measure a general set of expectations that the individual carries into new situations and his perception regarding his abilities to achieve goals in various situations and overcome challenges
The Screen for Child Anxiety Related Emotional Disorders (SCARED) | 3 months
  is a self-reported 41 questions scale for children and parents, designed to screen DSM-5 anxiety disorders
The Hebrew adaptation of The Children's Hope Scale (Snyder, 2002) | 3 months
  consists of 6 statements to which students respond on a 6-point Likert-type scale ranging from 1 (none of the time) to 6 (all of the time). There are three agency items (e.g., "I think I am doing pretty well") and three pathways items (e.g., "I can think of many ways to get things in life").
The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | 3 months
  a standardized, norm-referenced measure used by physical therapists and occupational therapists in clinic and school practice settings. It is an individually administered measure of fine and gross motor skills of children and youth, 4 through 21 years of age and is used by practitioners and researchers as a discriminative and evaluative measure to characterize motor performance, specifically in the areas of fine manual control, manual coordination, body coordination, and strength and agility.
The Short Sensory Profile (SSP) | 3 months
  The Short sensory profile (SSP; Dunn, 1999) is a 38- item questionnaire that assesses seven sensory domains: tactile, taste; smell; movement; under-responsive/seeks sensation; auditory filtering; low energy/weak, and visual/auditory
The Child Performance Skill Questionnaire (PSQ) | 3 months
  a questionnaire designed for parents to assess 3 skill domains: motor, process, and communication a questionnaire designed for parents to assess 3 skill domains: motor, process, and communication a questionnaire designed for parents to assess 3 skill domains: motor, process, and communication a questionnaire designed for parents to assess 3 skill domains: motor, process, and communication
The children Participation Questionnaire (CPQ) | 3 months
  a parent-reported questionnaire measuring participation of preschool children aged 4-6 years in their everyday activities
Canadian Occupational Performance Measure (COPM) (Law et al., 2014) | 3 months
  a standardized client-centered tool designed for use by occupational therapists to detect self-perceived change in occupational performance problems over time in children over the age of 5

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Helmer A, Delore E, Bart O. Horses and ADHD: the ASTride intervention for cognitive and emotional growth. Child Adolesc Psychiatry Ment Health. 2025 Nov 21;19(1):131. doi: 10.1186/s13034-025-00990-6. PMID 41272733